CLINICAL TRIAL: NCT01524458
Title: Prospective Study on the Feasibility and Effectiveness of Per-Oral Endoscopic Myotomy (P.O.E.M.) for Treatment of Primary Esophageal Motility Disorders
Acronym: POEM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Philip WY Chiu, Professor, Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2010.430
Record Dates: First submitted 2012-02-01; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2010-10

CONDITIONS: Primary Esophageal Motility Disorders Including Achalasia and Hypertensive LES

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- POEM (Experimental): To perform myotomy using endoscopy through a long submucosal tunnel
  Interventions: Procedure: Per-Oral Endoscopic Myotomy

INTERVENTIONS:
Procedure: Per-Oral Endoscopic Myotomy — To perform myotomy for lower esophageal sphincter using endoscope through a long submucosal tunnel

SUMMARY:
rimary spastic esophageal motility disorders, though uncommon, induce significant symptoms to patients including dysphagia, spastic chest pain, regurgitation as well as heartburn. The commonest causes of spastic esophageal motility disorders included Achalasia, hypertensive lower esophageal sphincter (LES), Nutcracker esophagus and Diffuse esophageal spasm (DES). Majority of these diseases were diagnosed by manometry. Achalasia is the most common primary esophageal motility disorder in which the LES failed to relax with increased pressure. Currently the standard treatment for Achalasia and spastic motility disorders is Laparoscopic Myotomy. The development of Natural Orifices Transluminal Endoscopic Surgery (N.O.T.E.S.) has lead to a new way to perform myotomy - Peroral Endoscopic Myotomy (P.O.E.M.). Basically, through mucosal incision, a submucosal tunnel is created after identification of the level of gastroesophageal junction. Myotomy will be performed with endoscopic instruments and the entrance site will be closed with clips.

ELIGIBILITY:
Inclusion Criteria:

* All patients with age ranged 18 to 85 who had primary esophageal motility disorders will be recruited. The primary motility disorders included: Achalasia, hypertensive LES, Nutcracker esophagus and Diffuse esophageal spasm.

Exclusion Criteria:

1. Pregnancy
2. Informed consent not available
3. Previous history of esophagectomy or mediastinal surgery
4. Previous history of endoscopic resection for early esophageal cancers, inclduing endoscopic mucosal resection and endsocopic submucosal dissection
5. End-stage Achalasia with dilated esophagus more than 6cm on Barium swllow

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2010-07

PRIMARY OUTCOMES:
Relief of Dysphagia | 4 weeks

SECONDARY OUTCOMES:
Complication | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip WY Chiu, MD, Principal Investigator — Dept of Surgery, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China